CLINICAL TRIAL: NCT02879890
Title: Impact of Comorbidities on Measure of Indirect Utility Change in Hip and Knee Ostearthritis
Brief Title: Comorbidities and Indirect Health State Utility in Hip and Knee Osteoarthritis
Acronym: COMUTAR
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: Comutar1
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
National cohort study aimed to investigate the impact of comorbidities (number and type of comorbidities) on health utility state change in lower lim osteoarthritis (hip and knee OA).

DETAILED DESCRIPTION:
The concept of health utility state was developed by economists to explain individual choices and preferences for health states. It is expressed as the "desirability or preference that individuals exhibit for the condition". This health utility state can be measured indirectly using health-relation quality of life questionnaires.

Chronic diseases such as OA are known to be associated with impairment of quality of life. Given that OA prevalence increases with age, OA is often associated with other diseases (comorbidities). A cross-sectional study showed that comorbidities are associated with lower health utility state in OA. Investigation of longitudinal impact of comorbidities on health utility state change is need.

Main objective: Determine the impact of comorbidities on change in health utility state among patients with lower limb OA.

Secondary objective: Determine the Minimal Clinically important Difference in health utility state among patients with lower limb OA.

The COMUTAR study uses longitudinal data from the Knee and Hip Osteoarthritis Longitudinal Assessment (KHOALA) cohort study. Health utility state is measured indirectly using Medical Outcome Study Short Form-36 quality of life questionnaire Comorbidities are assessed using the Functional Comorbidity Index

ELIGIBILITY:
Inclusion Criteria:

* age: 40-75 years
* Uni or bilateral lower limb osteoarthritis (OA) according to the American College of Rheumatology (ACR) and European league against rheumatism (EULAR) criteria

Exclusion Criteria:

* Hip or knee prothesis
* Antecedent of osteotomy
* Severe comorbidity
* Adult under legal protection

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population-based
Sampling Method: Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2009-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in health utility state | Five years
  Change in health state utility score between the inclusion in the KHOALA cohort and 5 years later (T5-T0)

SECONDARY OUTCOMES:
Minimal Clinically Important Difference (MCID) of health utility state | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Francis GUILLEMIN, MD, PhD, Principal Investigator — CHRU Nancy

IPD SHARING:
Plan to Share IPD: Yes
Open to partnership